CLINICAL TRIAL: NCT05424250
Title: Optimizing Exposure Therapy Via Occasional Aversive Imagery: A Randomized Controlled Trial With Spider Fearful Individuals
Brief Title: Optimizing Exposure Using Occasional Aversive Imagery in Spider Fearful Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPEX_SPIDER
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Spider Fear; Arachnophobia
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure + occasional aversive imagination (Experimental): repeated imaginations of the participants' most feared apprehension during extinction training with seven standardized exposure steps
  Interventions: Behavioral: occasional aversive imagination; Behavioral: Exposure
- Exposure (Active Comparator): Standard extinction training with seven standardized exposure steps
  Interventions: Behavioral: Exposure

INTERVENTIONS:
Behavioral: occasional aversive imagination — During six of the 27 exposure trials, participants in the experimental group are asked to imagine their most feared outcome towards spiders as vividly as possible while completing the specific trial.
  Arms: Exposure + occasional aversive imagination
Behavioral: Exposure — • All participants complete an exposure training session (approx. 75 min) with seven exposure steps, which are repeated between one and five times (e.g. Step 4: directing the spider with a pen by touching its legs at least five times per repetition; this step must be repeated five times before continuing to the next step). One repetition per step is considered one trial, therefore each participant aims to complete 27 exposure trials.

SUMMARY:
The effectiveness of an optimized extinction training is investigated in spider-fearful individuals. Participants will undergo a one-session standardized extinction training, either with or without occasional metal imagination of most feared apprehension towards spiders. The effectiveness of the training is measured by symptom improvement according to subjective ratings and behavioural avoidance tests one week later.

DETAILED DESCRIPTION:
The present study aims to investigate the applicability of an optimized exposure training using imagination. Exposure training is an effective approach to the treatment of various anxiety disorders. However, there are a significant number of patients who do not benefit or who develop anxiety following successful treatment. The process of extinction underlying exposure is the focus of current research on optimizing exposure. In this regard, one promising approach for improving extinction learning involves the occasional presentation of fear-generating stimuli (unconditioned stimuli [US]; often an electrical stimulus in experimental studies) during extinction (occasional reinforced extinction, ORE). Previous experimental studies provide preliminary evidence for a less pronounced return of fear after extinction training with occasional presentation of the US. In clinical practice, this strategy is recommended to optimize extinction learning in the treatment of individuals with anxiety. However, the transfer of the procedure used (real presentation of an unconditioned stimulus) into clinical practice seems difficult to realize. One way to facilitate the transfer of the ORE approach into clinical practice could be the use of vivid imagination of a personally relevant fear-generating situation during extinction training/exposure (e.g., patients' central concerns). Therefore, the aim of the present study is to examine the applicability of ORE using imagination. In this context, a standardized extinction training either with or without mental imagination of a personally relevant fear situation (e.g., central concern of the consequences when confronted with spiders) will be performed in individuals with spider-fearful individuals. The approach used for individuals with spider fear is well established and has been successfully implemented in previous studies by instructed trainers (e.g., individuals with a bachelor's degree in psychology). The aim of this randomized controlled trial in healthy individuals with increased fear of spiders is to investigate whether optimized extinction training (extinction training + imagination) is more effective in reducing fear of spiders in the long term compared to standard extinction training.

ELIGIBILITY:
Inclusion Criteria:

* Elevated score on Spider Phobia Questionnaire (SPQ) > 17

Exclusion Criteria:

* Severe allergies to bees/spiders/insects
* current psychotherapeutic/psychiatric treatment
* past psychotherapeutic/psychiatric treatment due to anxiety problems
* current or past psychotic symptoms
* current suicidal intent
* experience with exposure-based treatment
* current psychopharmacological medication
* severe cardiovascular, respiratory or neurological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Spider Phobia Questionnaire (SPQ) | Change from baseline to post-treatment (i.e., 7-9 days)
  31-item true/false questionnaire assessing symptoms of arachnophobia. Scores range from 0 to 31, with greater scores representing greater fear of spiders. Spider phobic individuals have obtained mean scores of 23.20 (SD = 2.90) and 23.76 (SD = 3.80) on the SPQ.
Behavioral Approach Test (BAT) | Change from baseline to post-treatment (i.e., 7-9 days)
  Number of test steps fully completed (0-14 steps)
Fear rating | Change from baseline to post-treatment (i.e., 7-9 days)
  Maximum fear rating on a scale from 0 (no fear) to 100 (severe fear) recorded once during BAT

SECONDARY OUTCOMES:
Fear of Spider Questionnaire (FSQ) | Change from baseline to post-treatment (i.e., 7-9 days)
  14-item questionnaire on a 7-point Likert scale (0 = 'I don't agree at all'; 6 = 'I completely agree') assessing symptoms of arachnophobia. Total score range: 0 to 84. Higher scores indicate worse severity of arachnophobia.
Change in anxiety sensitivity (ASI-3) | change from baseline to post-treatment (i.e. 7-9 days)
  The Anxiety Sensitivity Index (ASI-3) is a self-report measure of fear of anxiety-related body symptoms (i.e., anxiety sensitivity). Total score range: 0 to 72. Higher scores indicate worse anxiety sensitivity.
PROMIS Emotional Distress-Anxiety-Short Form | change from baseline to post-treatment (i.e. 7-9 days)
  The DSM-5-TR Level 2-Anxiety-Adult measure is the 7-item PROMIS Anxiety Short Form that assesses the pure domain of anxiety in individuals age 18 and older. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
US expectancy and fear ratings | Baseline
  Ratings of US expectancy and fear during exposure training on a scale from 0 (I don't expect my feared outcome/I am not scared at this moment) to 100 (I completely expect my feared outcome to happen/I am severely scared at this moment). Specifically, we asked participants to rate their US expectancy and fear before and during each of the 27 trials.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Benke, PhD, Principal Investigator — Philipps University Marburg; Christiane Pané-Farré, PhD, Principal Investigator — Philipps University Marburg; Dorothee Scheuermann, M.Sc., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University Marburg, Marburg, Hesse, Germany

REFERENCES:
- [Background] Craske MG, Treanor M, Conway CC, Zbozinek T, Vervliet B. Maximizing exposure therapy: an inhibitory learning approach. Behav Res Ther. 2014 Jul;58:10-23. doi: 10.1016/j.brat.2014.04.006. Epub 2014 May 9. PMID 24864005
- [Background] Culver NC, Stevens S, Fanselow MS, Craske MG. Building physiological toughness: Some aversive events during extinction may attenuate return of fear. J Behav Ther Exp Psychiatry. 2018 Mar;58:18-28. doi: 10.1016/j.jbtep.2017.07.003. Epub 2017 Jul 25. PMID 28777975
- [Background] Lipp OV, Ryan KM, Luck CC, Craske MG, Waters AM. Presentation of unpaired unconditional stimuli during extinction reduces renewal of conditional fear and slows re-acquisition. Psychophysiology. 2021 Oct;58(10):e13899. doi: 10.1111/psyp.13899. Epub 2021 Jul 6. PMID 34231228
- [Background] Shiban Y, Wittmann J, Weissinger M, Muhlberger A. Gradual extinction reduces reinstatement. Front Behav Neurosci. 2015 Sep 15;9:254. doi: 10.3389/fnbeh.2015.00254. eCollection 2015. PMID 26441581
- [Background] Thompson A, McEvoy PM, Lipp OV. Enhancing extinction learning: Occasional presentations of the unconditioned stimulus during extinction eliminate spontaneous recovery, but not necessarily reacquisition of fear. Behav Res Ther. 2018 Sep;108:29-39. doi: 10.1016/j.brat.2018.07.001. Epub 2018 Jul 3. PMID 29981936